CLINICAL TRIAL: NCT05129748
Title: A Multicenter Randomized Phase II Clinical Trial of the Efficacy of Sodium Thiosulfate and Mannitol in Reducing Ototoxicity in Adult Patients Receiving Cisplatin Chemotherapy
Brief Title: Efficacy of Sodium Thiosulfate and Mannitol in Reducing Ototoxicity in Adult Patients Receiving Cisplatin Chemotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1818
Record Dates: First submitted 2021-11-03; First posted 2021-11-22 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Ototoxic Hearing Loss
Keywords: Hearing Loss; Deafness; Cisplatin-induced Ototoxicity; Sensorineural hearing loss; Ear diseases; Sodium Thiosulfate
MeSH Terms: conditions — Hearing Loss; Deafness; Hearing Loss, Sensorineural; Ear Diseases | interventions — sodium thiosulfate; Mannitol

STUDY DESIGN:
Intervention Model Description: 1:1 randomization between cisplatin alone, and cisplatin, sodium thiosulfate and mannitol.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Cisplatin-based Chemotherapy + Sodium Thiosulfate + Mannitol (Experimental): Participants will receive the standard of care (cisplatin-based chemotherapy) plus the experimental treatment of Sodium Thiosulfate and Mannitol. Both drugs will be administered IV 4 - 8 hours following chemotherapy treatment, as part of post-chemotherapy hydration.
  Interventions: Drug: Sodium Thiosulfate + Mannitol
- Standard Cisplatin-based Chemotherapy (No Intervention): Participants will receive the standard of care (cisplatin-based chemotherapy) only.

INTERVENTIONS:
Drug: Sodium Thiosulfate + Mannitol — Drug delivery will be sequential, where Mannitol will be infused over 30 minutes and Sodium Thiosulfate will be infused over 15 minutes.
  Arms: Standard Cisplatin-based Chemotherapy + Sodium Thiosulfate + Mannitol

SUMMARY:
One common side effect of cisplatin chemotherapy is ototoxicity. The drugs sodium thiosulfate and mannitol may protect against cisplatin-induced hearing loss. Specifically, sodium thiosulfate has been found to protect the cells in the inner ear, and may therefore prevent hearing loss. Mannitol can help sodium thiosulfate enter the inner ear, and ponteially increase the effectiveness of sodium thiosulfate. This study aims to assess the efficacy of sodium thiosulfate and mannitol to reduce the hearing impairment caused by cisplatin chemotherapy.

DETAILED DESCRIPTION:
Randomized phase II clinical trial: with 1:1 randomization between cisplatin alone, and cisplatin + sodium thiosulfate and mannitol. Participants will first be recruited into a 2-year pilot feasibility study of 24 patients (12 in each arm). The pilot study will be performed to evaluate the feasibility of the trial as defined by the following factors: treatment outcomes, occurrence of adverse events, logistics of treatment delivery, as well as dropout and recruitment rates. The results from the pilot study will support the safety, efficacy, and effectiveness of the sodium thiosuldate and mannitol treatment, confirm feasibility using the factors mentioned above, and serve as an earlier-phase developmental function to enhance the probability of success of the subsequent clinical trial. Participants will complete various pre-treatment hearing tests. Participants will receive sodium thiosulfate and mannitol 4 - 8 hours following chemotherapy treatment. The control group will not receive the experimental intervention. Follow-up hearing tests will be performed at select time intervals following completion of their cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients undertaking systemic cisplatin therapy as part of their cancer treatment
* Age ≥ 18
* Willing to provide informed consent
* ECOG performance status 0-2
* For female of child-bearing potential, a negative pregnancy test (beta-HCG) prior to study treatment is required
* Any patient who is of reproductive age should provide written agreement to use adequate contraception for the duration of the trial

Exclusion Criteria:

* Age less than 18
* Preexisting severe to profound sensorineural hearing loss (unilateral or bilateral) (speech reception threshold >70dB, or word recognition score <50%) as confirmed with an audiogram
* History of Meniere's or fluctuating hearing loss
* Asymmetrical hearing loss (bone conduction threshold difference of: (a) 20 dB threshold difference at a single frequency, (b) 15 dB threshold difference at 2 frequencies, (c) 10 dB threshold difference at 3 frequencies
* Abnormal renal function (creatinine clearance <60 ml/min)
* Abnormal liver function (liver function tests (ALT and ALP) >2.5 times upper limit of normal without liver metastasis and >5 times upper limit of normal with liver metastasis
* Previous hypersensitivity to STS or mannitol
* Pregnant and/or nursing women
* Patient unable to follow the protocol for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in hearing threshold with sodium thiosulfate and mannitol administration | 2 months
  The primary outcome measure of this study will be a comparison of hearing loss between the control and experimental groups. More specifically, each ear will be scored as having hearing loss if there is a greater than 10dB hearing loss in three contiguous frequencies. This will be measured via threshold hearing tests.

SECONDARY OUTCOMES:
To monitor potential oncological impact of sodium thiosulfate and mannitol on long-term renal clearance | 12 months
  Participants will be monitored for renal function via serum creatinine (umol/L) and creatinine clearance (ml/min).
To monitor potential oncological impact of sodium thiosulfate and mannitol on disease free survival | 12 months
  Participants will be monitored for disease free survival via cancer staging details and clinical prognosis
To monitor potential oncological impact of sodium thiosulfate and mannitol on overall survival | 12 months
  Participants will be monitored for overall survival via time in months
To assess the short and long-term adverse event reporting from combination of sodium thiosulfate, mannitol and cisplatin. | 12 months
  To determine the causality of adverse events and serious adverse events and grading according to National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v.5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No